CLINICAL TRIAL: NCT04367467
Title: Effect of PARP Inhibitors on Glomerular Filtration Rate
Status: Terminated | Type: Observational
Why Stopped: Due to constraints of COVID19, we were unable to recruit on-site for this study.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 829785
Record Dates: First submitted 2020-04-03; First posted 2020-04-29 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor; Ovarian Cancer; Breast Cancer
Keywords: PARPi; Kidney function; Cystatin-C
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Kidney function will be assessed by serum creatinine, serum cystatin C, and urine creatinine clearance calculation for patients who opt-in to 24 hour urine collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with solid tumors receiving PARPi: Kidney function will be assessed by serum creatinine, serum cystatin C, and urine creatinine clearance calculation for patients who opt-in to 24 hour urine collection.
  These laboratory measures will be completed by patients at the following time points:
  * Timepoint A: Baseline (prior to PARP inhibitor initiation, at the time of standard of care clinical testing)
  * Timepoint B: On-treatment (within 3-9 weeks of PARP inhibitor initiation, at the time of standard of care clinical testing)
  * Timepoint C: Post-treatment (within 4 weeks of PARP inhibitor discontinuation, only for those patients with clinically significant changes in GFR based on serum creatinine, cystatin C, or 24 hour urinalysis at Timepoint B
  Interventions: Other: Kidney Function Test

INTERVENTIONS:
Other: Kidney Function Test — Cystatin-C measurement

SUMMARY:
The purpose of this study is to observe whether PARP inhibitors have an effect on serum creatinine level, and whether this reflects a change in creatinine secretion or a true change in kidney function.

DETAILED DESCRIPTION:
PARPi medications interact with transporters along the renal tubules involved in the secretion of creatinine and an increase in serum creatinine is often observed in patients treated with these agents; however, it is not known whether PARP inhibitors are associated with an actual change in the glomerular filtration rate, or if the observed elevations of serum creatinine are a result of a drug effect on creatinine secretion unrelated to changes in kidney function. The investigators therefore propose a prospective observational study to examine the incidence of elevation in serum creatinine from baseline levels in patients initiated on PARP inhibitors and compare the estimated glomerular filtration rate based on creatinine to that from alternative tests.

The primary purposes of this study are to:

* Assess the incidence of increase in serum creatinine in patients with a solid-organ cancer on treatment with a PARP inhibitor.
* To compare the estimated glomerular filtration rate based on serum creatinine with that of alternative biomarkers to assess whether changes in serum creatinine reflect changes in kidney function or creatinine secretion.
* To examine the persistence or resolution of creatinine increase and/or GFR decrease noted after discontinuation of PARPi

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 years or older
* Diagnosed with any solid organ cancer
* Planned to receive a PARP inhibitor (olaparib, niraparib, rucaparib, veliparib, or talazoparib)
* Able to consent to study related procedures
* If unable to give informed consent, must have healthcare proxy or legally authorized representative
* Fluent in conversational English (Informed Consent form currently in English language)

Exclusion Criteria:

* Patients who will not receive ongoing cancer care at Penn Medicine
* Major psychiatric illness or cognitive impairment that in the judgment of the study investigators or study staff would preclude study participation
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff
* Patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited from the medical and gynecologic oncology practices at the Abramson Cancer Center / University of Pennsylvania. Patients that are 18+ years or older with a solid organ cancer who are being initiated on PARP inhibitor therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in eGFR from Baseline to On-Treatment, 3-9 weeks after PARPi Initiation (Time Point B) | Study labs will be obtained within 3-9 weeks after PARPi is initiated
  Change in eGFR from baselineto on-treatment by ≥20% as measured using either cystatin C or 24h urine collection

SECONDARY OUTCOMES:
Within 4 Weeks of Post-discontinuation of PARPi (Time Point C) for patients with clinically significant changes in eGFR based on serum creatinine, cystatin C, or 24 hour urinalysis at Timepoint B | Post-treatment (within 4 weeks of PARP inhibitor discontinuation, only for those patients with clinically significant changes in GFR based on serum creatinine, cystatin C, or 24 hour urinalysis at Timepoint B
  The percentage of patients who experience a eGFR reduction of ≥30%, and/or

CONTACTS AND LOCATIONS:
Overall Officials: Payal Shah, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No